CLINICAL TRIAL: NCT03745664
Title: Effect of Corticosteroids On MyocardiaL Injury Among Patients Hospitalized for Community-AcquirEd PneUMonia - COLOSSEUM TRIAL
Brief Title: Corticosteroids and Myocardial Injury in CAP (COLOSSEUM TRIAL)
Acronym: COLOSSEUM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Francesco Violi, Prof. Francesco Violi, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COLOSSEUM trial - Rif 5133
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Community-acquired Pneumonia
Keywords: corticosteroids
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Methylprednisolone Hemisuccinate; Saline Solution; Injections

STUDY DESIGN:
Intervention Model Description: Phase 3, multicenter, double-blind, placebo-controlled, randomized, intervention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Doctors, staff and any primary care provider/s involved in the participant's non-trial management will be blinded to the group allocations. Individual participants will be not told their group allocation until the end of their involvement in the trial and after the completion of the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Methylprednisolone Sodium Succinate (20mg/ml) will be given at the dose of 40 mg/day (20 mg x 2/day).
  The treatment will last 7 days (or the time of hospitalization if the patient is discharged in a period less or more than 7 days).
  Interventions: Drug: Methylprednisolone Sodium Succinate
- Placebo group (Placebo Comparator): Saline Solution for Injection will be given ath the dose of 2 ml/day. The treatment placebo will last 7 days (or the time of hospitalization if the patient is discharged in a period less or more than 7 days).
  Interventions: Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Methylprednisolone Sodium Succinate — During hospitalization, 40 mg of methylprednisolone (20 mg/ml) will be given intravenously twice a day (20 mg every 12 hours).
  Arms: Treatment group
Drug: Saline Solution for Injection — During hospitalization, 2 ml of Saline Solution for Injection will be given intravenously twice a day (2 ml every 12 hours).
  Arms: Placebo group

SUMMARY:
Community-acquired pneumonia (CAP) is often complicated by elevation of cardiac troponin, a marker of myocardial injury, that can be isolated or associated to myocardial infarction (MI). A retrospective study showed that corticosteroid treatment lowers incidence of MI during the hospital-stay.

The aim of this clinical trial is to examine whether in-hospital treatment with iv methylprednisolone (20 mg b.i.d) may reduce myocardial injury, as assessed by serum high-sensitivity cardiac T Troponin) and eventually cardiovascular events during a short- and long-term follow-up in patients hospitalized CAP.

DETAILED DESCRIPTION:
Background. Community-acquired pneumonia (CAP) is often complicated by elevation of cardiac troponin, a marker of myocardial injury, that can be isolated or associated to myocardial infarction (MI). A retrospective study showed that corticosteroid treatment lowers incidence of MI during the hospital-stay. No data exist so far on the effect of corticosteroids on myocardial injury in CAP patients.

Study design. Double-blind randomized placebo-controlled trial. One hundred twenty-two eligible patients will be randomized to a week treatment with iv methylprednisolone (20 mg b.i.d) or placebo from hospital admission. Serum hs-cTnT will be measured at admission and every day until up 3 days from admission. ECG will be monitored every day until discharge. After dismission, all patients will be followed-up 2 years.

Aims of the study. Primary objective of the study is to evaluate if methylprednisolone is able to reduce myocardial injury, as assessed by serum high-sensitivity cardiac T Troponin (hs-cTnT), in a cohort of patients hospitalized for CAP.

Secondary aims are to evaluate the potential effect of methylprednisolone on cardiovascular events during hospitalization, at 30 day from hospital admission and during 2 years' follow-up. The trial will also examine whether the potential protective effects of methylprednisolone might be due to platelet activation down-regulation.

ELIGIBILITY:
Inclusion Criteria:

Hospitalization for community-acquired pneumonia

Exclusion Criteria:

1. Use of corticosteroids in the previous 30 days
2. Health Care-Associated Pneumonia
3. Reported severe immunosuppression (human immunodeficiency virus infection, immunosuppressive conditions or medications)
4. Preexisting medical condition with a life expectancy of less than 3 months
5. Uncontrolled diabetes mellitus
6. Gastritis with or without major gastrointestinal bleeding within 3 months
7. Any condition requiring acute treatment with glucocorticoids

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-05-16 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
High sensitivity cardiac T troponin (myocardial injury biomarker) | 7 days
  Primary endpoint of the study will be a significant reduction of hs-cTnT increase. Hs-cTnT will be measured . Hs-cTnT levels will be measured by the Elecsys 2010 (Roche Diagnostics, Indianapolis, IN) in a dedicated core laboratory.

SECONDARY OUTCOMES:
Serum TxB2 (biomarker of platelet activation) | 7 days
  Serum Thromboxane (Tx) B2 will be measured on blood samples obtained at admission, after 72 hours and at hospital discharge (within 7 days).
sP-selectin (biomarker of platelet activation). | 7 days
  Plasma sP-selectin will be measured on blood samples obtained at admission, after 72 hours and at hospital discharge (within 7 days).
sCD40L (biomarker of platelet activation). | 7 days
  Plasma sCD40L will be measured on blood sample obtained at admission, after 72 hours and at hospital discharge (within 7 days).
High-sensitivity C-Reactive Protein | 7 days
  Serum high-sensitivity C-Reactive Protein will be measured in blood samples obtained at admission, after 72 hours and at hospital discharge (within 7 days).
Serum sNOX2-dp (biomarker of oxidative stress) | 7 days
  Serum sNOX2-dp will be measured on blood samples obtained at admission, after 72 hours and at hospital discharge (within 7 days). Blood levels of soluble NOX2-derived peptide (sNOX2-dp), a marker of NADPH oxidase activation, will be detected by ELISA as previously described (Pignatelli P et al Arterioscler Thromb Vasc Biol 2010;30:360-7).
Serum F2-isoprostanes (biomarker of oxidative stress) | 7 days
  Serum F2-isoprostane (8-iso-PGF2α -III) will be measured by the enzyme immunoassay method in blood samples obtained at admission, after 72 horus and at hospital discharge (within 7 days).
Urinary F2-isoprostanes (biomarker of oxidative stress) | 7 days
  F2-isoprostanes will be measured in urine samples collected at admission, after 72 horus and at hospital discharge (within 7 days).
Cardiovascular events during hospitalization. | 7 days
  This composite outcome will consist in any of the following events during hospitalization: acute myocardial infarction, new or worsening heart failure, new onset atrial fibrillation, stroke, cardiovascular death.
Major adverse cardiac and cerebrovascular events (MACCE) at 30 days. | 30 days
  This composite outcome will consist in any of the following events during a 30-days follow-up: cardiovascular death, myocardial infarction and stroke.
Major adverse cardiac and cerebrovascular events (MACCE) during a a long-term follow-up. | 2 years
  This composite outcome will consist in any of the following events during a 2-years f follow-up: cardiovascular death, myocardial infarction and stroke.
Short-term mortality | 30 days
  Death for any cause during a 30-days follow-up
Long-term mortality | 2 years
  Death for any cause during a2 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — University of Roma La Sapienza; Roberto Cangemi, Study Director — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cangemi R, Casciaro M, Rossi E, Calvieri C, Bucci T, Calabrese CM, Taliani G, Falcone M, Palange P, Bertazzoni G, Farcomeni A, Grieco S, Pignatelli P, Violi F; SIXTUS Study Group; SIXTUS Study Group. Platelet activation is associated with myocardial infarction in patients with pneumonia. J Am Coll Cardiol. 2014 Nov 4;64(18):1917-25. doi: 10.1016/j.jacc.2014.07.985. Epub 2014 Oct 27. PMID 25444147
- [Background] Cangemi R, Falcone M, Taliani G, Calvieri C, Tiseo G, Romiti GF, Bertazzoni G, Farcomeni A, Violi F; SIXTUS Study Group. Corticosteroid Use and Incident Myocardial Infarction in Adults Hospitalized for Community-acquired Pneumonia. Ann Am Thorac Soc. 2019 Jan;16(1):91-98. doi: 10.1513/AnnalsATS.201806-419OC. PMID 30188173
- [Background] Cangemi R, Carnevale R, Nocella C, Calvieri C, Cammisotto V, Novo M, Castellani V, D'Amico A, Zerbinati C, Stefanini L, Violi F; SIXTUS Study Group. Glucocorticoids impair platelet thromboxane biosynthesis in community-acquired pneumonia. Pharmacol Res. 2018 May;131:66-74. doi: 10.1016/j.phrs.2018.03.014. Epub 2018 Mar 22. PMID 29577968
- [Background] Liverani E, Banerjee S, Roberts W, Naseem KM, Perretti M. Prednisolone exerts exquisite inhibitory properties on platelet functions. Biochem Pharmacol. 2012 May 15;83(10):1364-73. doi: 10.1016/j.bcp.2012.02.006. Epub 2012 Feb 16. PMID 22366284